CLINICAL TRIAL: NCT00789646
Title: Painless Subconjunctival Antibiotic and Antifungal Injection in Corneal Ulcer Patients.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Very slow in enrolling participants
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Pramote Euasobhon, Dr, Mahidol University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SI 271/2008
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Corneal Ulcer
Keywords: corneal ulcer; painless; subconjunctival injection; antibiotics; antifungal; lidocaine
MeSH Terms: conditions — Corneal Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NSS/Lidocaine (Experimental): First injection: Normal saline Second injection: 2% Lidocaine without adrenaline
  Interventions: Procedure: NSS/Lidocaine
- Lidocaine/NSS (Experimental): First injection: 2% Lidocaine without adrenaline Second injection: Normal saline
  Interventions: Procedure: Lidocaine/NSS

INTERVENTIONS:
Procedure: Lidocaine/NSS — First injection: subconjunctival 2% lidocaine without adrenaline 0.4 ml. before antibiotic injection Second injection (24 hours later): subconjunctival NSS 0.4 ml. before antibiotic injection
  Arms: Lidocaine/NSS
Procedure: NSS/Lidocaine — First injection: subconjunctival NSS 0.4 ml. before antibiotic injection Second injection (24 hours later): subconjunctival 2% lidocaine without adrenaline 0.4 ml. before antibiotic injection
  Arms: NSS/Lidocaine

SUMMARY:
The propose of this study is to determine the efficacy of 2% xylocaine in reducing pain due to subconjunctival antibiotic and antifungal injection.

ELIGIBILITY:
Inclusion Criteria:

* The corneal ulcer patients who are diagnosed by ophthalmologist and have 2 of 3 in these following features.

  1. corneal epithelial defect with stromal infiltration
  2. reaction in anterior chamber
  3. positive for bacteria or fungus
* The patients have to receive subconjunctival antibiotic injection twice at least.
* The patients must be informed consent.

Exclusion Criteria:

* The patients who have history of allergy of local anesthetics, antibiotics or antifungal drugs.
* The patients who administered NSAIDs or weak opioids within 24 hours prior to subconjunctival antibiotic/antifungal injection.
* Unable to cooperate with the treatment.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Numeric rating scale | immediately after injection

SECONDARY OUTCOMES:
Side effects | 24 hours after injection